CLINICAL TRIAL: NCT02892474
Title: Hybrid Coronary Revascularization Versus Coronary Artery Bypass Surgery for Treatment of Multivessel Coronary Disease
Brief Title: HCR vs. CABG Study
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Michael Halkos, Associate Professor of Surgery, Emory University
Other Study IDs: IRB00089868
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Arteriosclerosis; Hybrid Coronary Revascularization; Coronary Artery Bypass Grafting
MeSH Terms: conditions — Coronary Artery Disease | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hybrid Coronary Revascularization (HCR): Patients who are scheduled to have the hybrid coronary revascularization (HCR) procedure for treatment of multi-vessel coronary artery disease. The treatment plan is determined by the patient's doctor.
  Interventions: Procedure: Hybrid Coronary Revascularization (HCR)
- Coronary Artery Bypass Grafting (CABG): Patients who are scheduled to have the coronary artery bypass grafting (CABG) procedure for treatment of multi-vessel coronary artery disease. The treatment plan is determined by the patient's doctor.
  Interventions: Procedure: Coronary Artery Bypass Grafting (CABG)

INTERVENTIONS:
Procedure: Hybrid Coronary Revascularization (HCR) — Hybrid coronary revascularization (HCR) is a combination of surgery and catheter procedures to open up clogged heart arteries. HCR is the intentional combination of coronary artery bypass grafting (CABG) and percutaneous coronary intervention (PCI). The HCR strategy combines grafting of the left anterior descending artery (LAD) coronary artery using the left internal mammary artery (LIMA) with PCI of non-LAD coronary stenoses. Drug-eluting stents are substituted for saphenous vein grafts (SVG) for non-LAD coronary targets, and the surgical LIMA to LAD bypass is performed, ideally through a minimally invasive, limited access, sternal-sparing approach.
  Groups: Hybrid Coronary Revascularization (HCR)
Procedure: Coronary Artery Bypass Grafting (CABG) — Coronary artery bypass grafting (CABG) is a surgery to create a new path for blood flow to the heart. A healthy section of vein or artery from elsewhere in the patient's body will be attached to the coronary artery just above and below the area of concern, to create a way for blood to bypass the blocked part of the coronary artery.
  Groups: Coronary Artery Bypass Grafting (CABG)

SUMMARY:
The purpose of the study is to find out if hybrid coronary revascularization (HCR) and coronary artery bypass grafting (CABG) procedure outcomes are similar. HCR is a combination of surgery and catheter procedures to open up clogged heart arteries. CABG is a surgical procedure to open up clogged heart arteries.

DETAILED DESCRIPTION:
Currently, it is not clear how the outcomes of hybrid coronary revascularization (HCR) compare with other treatments. The purpose of the study is to find out if HCR and coronary artery bypass grafting (CABG) procedure outcomes are similar. HCR is a combination of surgery and catheter procedures to open up clogged heart arteries. CABG is a surgical procedure to open up clogged heart arteries.

This study will collect information about the medical care participants receive during their planned procedure. No new testing or procedures will be done. Participants will have only the tests or procedures already planned by their doctor. The investigators will look at how well participants do after the procedure by assessing the outcomes of interest 30 days after surgery and, potentially, one year after surgery (funding dependent).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent
* Have multi-vessel coronary artery disease (CAD) involving the Left Anterior Descending (LAD) artery
* Have a clinical indication for revascularization
* Are a candidate for either HCR or CABG or both
* Anatomy suitable for HCR shall include

  1. Multi-vessel CAD involving the LAD and/or
  2. LAD disease and involvement of a major diagonal artery, both of which require revascularization

Exclusion Criteria:

* Prior cardiac operations
* Severe left ventricular dysfunction with ejection fraction (EF) < 30%
* Patients with chest radiation
* Body mass index (BMI) > 35
* Severe peripheral vascular disease (PVD)
* Acute ischemia requiring emergent traditional coronary artery bypass graft (CABG)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patient population for this trial consists of adult patients with multi-vessel coronary artery disease who are being treated with either hybrid coronary revascularization (HCR) or coronary artery bypass grafting (CABG), as determined by their doctor.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-07-27 (Actual); Study Completion 2018-07-27 (Actual)

PRIMARY OUTCOMES:
Comparison of major adverse cardiac and cerebrovascular events (MACCE) between groups | Up to one year
  Major adverse cardiac and cerebrovascular events (MACCE) will be assessed at 30 days and at one year after the index procedure. For the purpose of this trial, the components of MACCE include (1) all-cause mortality, (2) repeat revascularization, (3) stroke, and (4) myocardial infarction.

SECONDARY OUTCOMES:
Comparison of all-cause mortality between groups | Up to one year
  All-cause mortality will be assessed at 30 days and at one year after the index procedure.
Comparison of repeat revascularization between groups | Up to one year
  Repeat revascularization (all-cause) will be assessed at 30 days and at one year after the index procedure.
Comparison of stroke between groups | Up to one year
  The incidence and severity of strokes experienced between the groups will be assessed at 30 days and at one year after the index procedure, using the NIH Stroke Scale (NIHSS). The NIHSS is a 15-item neurologic examination stroke scale used to evaluate the effect of acute cerebral infarction on the levels of consciousness, language, neglect, visual-field loss, extraocular movement, motor strength, ataxia, dysarthria, and sensory loss. A trained observer rates the patent's ability to answer questions and perform activities. Ratings for each item are scored with 3 to 5 grades with 0 as normal, and there is an allowance for untestable items. The single patient assessment requires less than 10 minutes to complete.
Comparison of ischemia-driven repeat revascularization between groups | Up to one year
  The incidence of ischemia-driven revascularization experienced between the groups will be assessed at 30 days and at one year after the index procedure.
Comparison of ventilator time between groups | During hospitalization (typically 3-8 days)
  The amount of time each patient spends on a ventilator during the index hospitalization will be collected.
Comparison of surgical re-exploration between groups | During hospitalization (typically 3-8 days)
  The incidence of re-exploration due to postoperative bleeding will be collected during the index hospitalization.
Comparison of chest tube drainage complications between groups | During hospitalization (typically 3-8 days)
  Chest tube drainage complications will be collected during the index hospitalization.
Comparison of hospital length of stay between groups | During hospitalization (typically 3-8 days)
  Hospital length of stay will be collected during the index hospitalization.
Comparison of wound infection between groups | During hospitalization (typically 3-8 days)
  The incidence of wound infection will be collected during the index hospitalization.
Comparison of atrial fibrillation between groups | During hospitalization (typically 3-8 days)
  The incidence of atrial fibrillation will be collected during the index hospitalization.
Comparison of blood transfusion between groups | During hospitalization (typically 3-8 days)
  The incidence of blood transfusions will be collected during the index hospitalization.
Comparison of hospital readmission between groups | Up to one year
  Hospital readmission (all-cause and cardiac) will be assessed at 30 days and at one year after the index procedure.
Comparison of Angina Score between groups | Up to one year
  Angina will be assessed at Baseline (prior to surgery), 30 days after the procedure, and at one year after the index procedure.
  The Canadian Cardiovascular Society Angina Grading Scale will be used to categorize angina:
  * Class I - Ordinary physical activity does not cause angina, such as walking and climbing stairs. Angina with strenuous or rapid or prolonged exertion at work or recreation
  * Class II - Slight limitation of ordinary activity. Walking or climbing stairs rapidly, walking uphill, walking or stair climbing after meals, or in cold, or in wind, or under emotional stress or only during the few hours after awakening
  * Class III - Marked limitation of ordinary physical activity. Walking one or two blocks on the level and climbing one flight of stairs in normal conditions and at normal pace
  * Class IV - Inability to carry on a physical activity without discomfort - angina syndrome may be present at rest
Comparison of Duke Activity Scale Index (DASI) scores between groups | Up to one year
  The Duke Activity Scale Index (DASI) will be administered at Baseline (prior to surgery), 30 days after the procedure, and at one year after the index procedure. The DASI is a 12 item survey that asks about a patient's functional capacity in order to estimate peak oxygen uptake. Respondents answer "yes" or "no" to questions about their ability to do activities of different intensity levels.
Comparison of EuroQol EQ-5D scores between groups | Up to one year
  The EuroQol EQ-5D will be administered at Baseline (prior to surgery), 30 days after the procedure, and at one year after the index procedure. The EuroQol EQ-5D is a 6 item survey that asks about how a patient is feeling on the day of the survey in terms of mobility, self-care, usual activities, pain/discomfort, anxiety/depression, and how they rate their health on a scale of 0 to 100 (where 0 is the worst health imaginable and 100 is the best health imaginable).

CONTACTS AND LOCATIONS:
Overall Officials: Michael Halkos, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital Midtown, Atlanta, Georgia, United States